CLINICAL TRIAL: NCT03340649
Title: The Predictive Value of Hepatocyte Growth Factor and Soluble Receptor s-Met in Evaluating Sepsis Patient's Disease Severity and Prognosis
Brief Title: The Predictive Value of Hepatocyte Growth Factor and Soluble Receptor s-Met in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jingyuan,Xu (Other)
Responsible Party: Sponsor-Investigator, Jingyuan,Xu, Attending doctor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 2017ZDSYLL095-P01
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: taking peripheral blood — taking peripheral blood of no more than 3ml

SUMMARY:
To observe the changes of plasma hepatocyte growth factor and soluble receptor s-Met levels in patients with sepsis, and to explore its clinical significance.

DETAILED DESCRIPTION:
90 patients who diagnosed as sepsis were included in this study. Then keep blood samples from these patients in the first day, the third day, detect the hepatocyte growth factor and soluble receptor s-Met level in plasma byenzyme-linked immuno sorbent assay. Record Severity of illness and survival status of every patient within 28 days. Objective to evaluate the correlation between the level of hepatocyte growth factor and soluble receptor s-Met in plasma and the prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to ICU diagnosed of sepsis(sepsis3.0 criteria)
2. Patients signing informed consent

Exclusion Criteria:

1. Age is less than 18 years old or more than 80 years old
2. Pregnant women
3. Patients with tumor、hepatitis、liver cirrhosis、acute myocardial infarction、chronic renal tubular nephritis、interstitial pneumonia、acute pancreatitis、systemic lupus erythenatosus、ulcerative colitis、crohn's disease、HELLP syndrome
4. Prothrombin time is extension in patients with after liver transplantation
5. Patients with chronic renal failure
6. Patients after kidney transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sepsis patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-11-09 (Estimated); Primary Completion 2017-11-09 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 28-day
  28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: yi yang, doctor, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
no share IPD